CLINICAL TRIAL: NCT06003556
Title: PSMA-Guided Ablation of the Prostate: A Multicenter Randomized Controlled Trial
Brief Title: PSMA-Guided Ablation of the Prostate
Acronym: P-GAP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HREBA.CC-23-0330
Record Dates: First submitted 2023-08-07; First posted 2023-08-22 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Localized Prostate Carcinoma
Keywords: Prostate Cancer; PSMA Pet; Focal Therapy; Localized Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radionuclide Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSMA PET (Experimental): These patients will have been diagnosed with unilateral prostate cancer by standard of care diagnostic tests deemed eligible and interested in focal therapy. These patients will be randomized to undergo a single [18]F-PSMA-1007 PET/CT or PET/MRI scan prior to focal therapy. If they are diagnosed with bilateral disease, they will be ineligible for focal therapy and be referred for radical therapy. Those with unilateral disease will then proceed to focal therapy. They will then receive PSMA PET, MRI, and combined targeted and systematic biopsy 12 months after ablation
  Intravenous bolus injection of 4 MBq/kg +/- 10% of [18]F-PSMA-1007, up to a maximum of 400 MBq.
  Interventions: Diagnostic Test: PSMA-1007 Positron Emission Tomography (PET) scan
- No Additional Imaging (No Intervention): These patients will have been diagnosed with unilateral prostate cancer by standard of care diagnostic tests deemed eligible and interested in focal therapy. These patients will undergo no further testing and will undergo focal therapy.
  They will then receive PSMA PET, MRI, and combined targeted and systematic biopsy 12 months after ablation.
  Intravenous bolus injection of 4 MBq/kg +/- 10% of [18]F-PSMA-1007, up to a maximum of 400 MBq.

INTERVENTIONS:
Diagnostic Test: PSMA-1007 Positron Emission Tomography (PET) scan — Additional staging PET scan prior to focal therapy to focal therapy.
  Arms: PSMA PET

SUMMARY:
The goal of this phase 2 multicenter randomized controlled trial is to study the accuracy of second generation prostate specific membrane antigen (PSMA) positron emission tomography (PET; utilizing 18F-PSMA-1007) compared to standard of care multiparametric MRI and MRI targeted-prostate biopsy for staging in patients diagnosed with unilateral prostate cancer who are eligible for focal therapy.

The main question it aims to answer is:

Can PSMA PET improve diagnostic accuracy for the primary staging of Prostate Cancer for patients undergoing focal therapy thereby reducing residual and recurrence disease?

Participants who are eligible by current standard of care diagnostic workup will undergo 1:1 randomization to PSMA PET scan or no further imaging. Those diagnosed with bilateral disease by PSMA PET will be ineligible for focal therapy and be referred for radical therapy. Men with unilateral disease on PSMA PET and those randomized to no further imaging will then undergo focal therapy. All men undergoing focal therapy will receive PSMA PET, MRI, and combined targeted and systematic biopsy 12 months after ablation. The primary outcome will be the detection of Gleason Grade Group 2 or higher prostate cancer in men 12 months after hemigland ablation.

DETAILED DESCRIPTION:
1. Background & Rationale

   Focal therapy is emerging as a new treatment strategy for appropriately selected men with localized prostate cancer. Focal therapy (also called partial gland ablation) is the concept of treating only where the tumor is believed to be located within the prostate, leaving normal healthy regions of the prostate untreated. Thus, focal therapy minimizes treatment side effects such as erectile dysfunction and incontinence, while providing good cancer control.

   The foundation of performing oncologically sound partial gland ablation is possessing a high degree of diagnostic certainty that the tumor is limited to the region that is being treated and is not unknowingly present elsewhere in the gland. However, this is currently a major diagnostic challenge. The current diagnostic strategy for work-up of a patient for focal therapy is based on a pre-operative multiparametric MRI and combined targeted and systematic prostate biopsy showing intermediate risk prostate cancer localized to only one side of the prostate gland. This combination has been shown to accurately diagnose the final tumor grade in 96.5% of men. However, whole mount pathology data after radical prostatectomy shows that over 50% of cases that would pre-operatively have been deemed appropriate for focal therapy, which is a unilateral treatment, in fact harbour bilateral disease, which would mean that contralateral tumor would be inadvertently left untreated. Similarly, our group has shown that of the 35% of men who were found to have residual tumor after hemigland ablation of their prostate for unilateral disease, two-thirds of residual tumors were identified on the side contralateral to the ablative treatment. Therefore, our current gold standard pre-operative imaging and biopsy techniques are under staging many men who are undergoing focal therapy and a new paradigm is required to advance focal ablative treatments.

   PSMA PET is a new imaging technique that uses a radioligand that binds to prostate specific membrane antigen (PSMA). PSMA is expressed at high levels in prostate cancer and the degree of expression correlates proportionately with tumor grade. A second generation PSMA PET radioligand, called 18F-PSMA-1007, has been used extensively at our site and possesses the key attributes of minimal urinary excretion, high resolution, and a half-life that as Gallium based radioligands. This makes 18F-PSMA-1007 an excellent candidate for improving the intraprostatic diagnostic accuracy of prostate cancer localization in patients considering focal therapy as a treatment option.
2. Research Question & Objectives

   Primary outcome:

   The primary outcome is the detection of any clinically significant prostate cancer (defined as greater than or equal to Gleason Grade Group 2) at MRI-guided combined targeted and systematic biopsy 12 months after hemigland ablation.

   Secondary outcomes:
   * the number of men found to have bilateral disease on PSMA PET prior to hemi-gland ablation
   * the number of men found to have bilateral disease on PSMA PET after hemi-gland ablation
   * the rate of contralateral Gleason Grade Group 2 or greater prostate cancer at 12-month biopsy
   * the rate of contralateral Gleason Grade Group 2 or greater prostate cancer at final pathology in men undergoing radical prostatectomy after PSMA PET detected bilateral disease
   * 5-year failure free survival defined as freedom from radical or systematic therapies, metastasis, prostate cancer specific and overall survivals.
   * side effects of PSMA PET imaging
   * health economics analysis of PSMA PET prior to hemigland ablation
   * Quality of life outcomes will be assessed with validated questionnaires
3. Methods The investigators propose a multi-centre phase II randomized-controlled trial of 138 patients deemed appropriate for focal therapy based on current standard-of-care (SOC) diagnostic work-up to be randomized to receive 18F-PSMA-1007 imaging or no further imaging. Patients found to have bilateral disease by PSMA PET will be ineligible for focal therapy and will proceed with SOC treatments (radical prostatectomy or radiation therapy). Men with unilateral disease on PSMA PET as well as all men receiving no further imaging will undergo hemigland ablation followed by PSMA PET, MRI, and combined targeted and systematic biopsy 12 months after ablation. The primary outcome will be the detection of Gleason Grade Group 2 or higher prostate cancer in men 12 months after hemigland ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50
2. Clinical stage < T2b
3. PSA < 15
4. Combined targeted and systematic MRI-guided biopsy shows unilateral Gleason Grade Group 2 or 3 prostate cancer

Exclusion Criteria:

1. Unable to obtain consent
2. Weight >250 kg (weight limitation of scanners)
3. Unable to lie flat for 30 minutes to complete the PET imaging
4. Lack of intravenous access
5. eGFR < 40 mL/min/1.73 m2 and/or a history of a severe reaction to CT contrast
6. Prior androgen deprivation therapy or radiation therapy to prostate gland

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2029-02-26 (Estimated); Study Completion 2029-02-26 (Estimated)

PRIMARY OUTCOMES:
Tumor Staging- Detection of any clinically significant prostate cancer | 12 months after hemigland ablation.
  Detection of any clinically significant prostate cancer (defined as greater than or equal to Gleason Grade Group 2) at MRI-guided combined targeted and systematic biopsy

SECONDARY OUTCOMES:
Tumor Staging - bilateral disease on PSMA PET prior to hemi-gland ablation | Prior to hemigland ablation - at study enrollment
  The number of men found to have bilateral disease on PSMA PET prior to hemi-gland ablation
Tumor Staging - bilateral disease on PSMA PET after hemi-gland ablation | 12 months after hemigland ablation.
  The number of men found to have bilateral disease on PSMA PET after hemi-gland ablation
Tumor Staging- rate of contralateral Gleason Grade Group 2 or greater prostate cancer at biopsy | 12 months after hemigland ablation.
  The rate of contralateral Gleason Grade Group 2 or greater prostate cancer at time of biopsy
Tumor Staging - rate of contralateral Gleason Grade Group 2 or greater prostate cancer at final pathology | Through study completion, expected within 1 year of randomization
  The rate of contralateral Gleason Grade Group 2 or greater prostate cancer at final pathology in men undergoing radical prostatectomy after PSMA PET detected bilateral disease
Tumor Staging - 5-year failure free survival | 5 years after hemigland ablation
  5-year failure free survival defined as freedom from radical or systematic therapies, metastasis, prostate cancer specific and overall survivals.
Side Effects of Intervention | Immediately after the imaging
  Number of patients with Side effects of PSMA PET imaging
Early Economic analysis | 12 months after hemigland ablation
  Comparison of the direct health care system costs incurred by each patient in both trials arms at the 1 year mark after hemigland ablation. Health system resource utilisation data will be captured using the administrative data infrastructures of the health care systems hosting the study centres, combined with data from the study clinical case report form. Unit costs for all resources will be obtained from CIHI and health system specific cost databases.
Post Trial Economic analysis | Through Study Completion, completion by end of study at 5 year mark
  Comparison of the direct health care system costs incurred by each patient in both trials arms at the 5 year mark after hemigland ablation at the time of study completion. Health system resource utilisation data will be captured using the administrative data infrastructures of the health care systems hosting the study centres, combined with data from the study clinical case report form. Unit costs for all resources will be obtained from CIHI and health system specific cost databases.
Quality of Life Outcomes - EPIC-26 | Through Study Completion, completion by end of study at 5 year mark. Every 3 months for first year and every 6months-1 year after
  The EPIC-26 is a short form questionnaire designed to measure Quality of Life (QOL) issues in patients with prostate cancer. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale with higher scores representing better Health Related QOL.
Quality of Life Outcomes - AUA Symptom Score | Through Study Completion, completion by end of study at 5 year mark. Every 3 months for first year and every 6months-1 year after
  The AUA Symptom Score evaluates impact and severity of urinary symptoms in patients with benign prostatic hyperplasia (BPH). The AUA Symptom Score ranges from 0 to 35, with higher scores indicating more severe symptoms.
Quality of Life Outcomes - IIEF 5 | Through Study Completion, completion by end of study at 5 year mark. Every 3 months for first year and every 6months-1 year after
  The IIEF-5 is a short form version of a patient-reported outcome measure to evaluate erectile dysfunction and other sexual problems in men. THE IIEF-5 scale ranges from 5-25 with a higher score indicating less severe symptoms.
Quality of Life Outcomes - EQ-5D-5L | Through Study Completion, completion by end of study at 5 year mark. Every 3 months for first year and every 6months-1 year after
  The EQ-5D-5L questionnaire is a self-assessed, health-related, quality of life questionnaire that measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The questionnaire can be used to derive a summary index score, which ranges from 0.000 (death) to 1.000 (perfect health).

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Prostate Cancer Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No